CLINICAL TRIAL: NCT05178407
Title: Effect of Household Use of Multiple Micronutrient-fortified Bouillon on Micronutrient Status Among Women and Children in Two Districts in the Northern Region of Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of Ghana (Other); Newcastle University (Other); Penn State University (Other); Helen Keller International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1837253
Record Dates: First submitted 2021-11-29; First posted 2022-01-05 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Vitamin A Deficiency; Iron-deficiency; Folate Deficiency; Vitamin B 12 Deficiency; Zinc Deficiency; Anemia
Keywords: Micronutrient, Food Fortification,
MeSH Terms: conditions — Vitamin A Deficiency; Anemia, Iron-Deficiency; Folic Acid Deficiency; Vitamin B 12 Deficiency; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The two study groups will receive different bouillon formulations in packaging that is identical except for the study group code. Linkage between the study group codes and bouillon formulations will be known only to the bouillon producer and independent codekeepers, and not to the investigators, data collection staff, or participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple micronutrient-fortified bouillon cube (Experimental): 10-gram shrimp-flavoured bouillon cube, fortified with 6 micronutrients
  Enrolled participants will receive a household bouillon ration for use in daily cooking (ad lib). Bouillon rations will be replenished every 2 weeks for the study duration of 38 weeks (non-pregnant, non-lactating women 15-49 y and children 2-5 y) or 12 weeks (lactating women 15-49 y and 4-18 mo postpartum).
  Interventions: Dietary Supplement: Multiple micronutrient-fortified bouillon cube
- Control bouillon cube (iodine only) (Placebo Comparator): 10-gram shrimp-flavoured bouillon cube, fortified with iodine
  Enrolled participants will receive a household bouillon ration for use in daily cooking (ad lib). Bouillon rations will be replenished every 2 weeks for the study duration of 38 weeks (non-pregnant, non-lactating women 15-49 y and children 2-5 y) or 12 weeks (lactating women 15-49 y and 4-18 mo postpartum).
  Interventions: Dietary Supplement: Control bouillon cube (iodine-only)

INTERVENTIONS:
Dietary Supplement: Multiple micronutrient-fortified bouillon cube — Bouillon cube fortified with 80 µg/g folic acid, 1.2 µg/g Vitamin B12, 3 mg/g Zinc (ZnO), 4 mg/g Iron (FePP/citric acid/trisodium citrate), 200 µg/g Vitamin A (retinyl palmitate), 30 µg/g Iodine (KIO3)
  Arms: Multiple micronutrient-fortified bouillon cube
Dietary Supplement: Control bouillon cube (iodine-only) — Bouillon cube fortified with 30 µg/g Iodine (KIO3)
  Arms: Control bouillon cube (iodine only)

SUMMARY:
Background: Micronutrient (MN) deficiencies are severe and widespread in West Africa, particularly among young children and women of reproductive age. Bouillon is a promising food fortification vehicle because the product is centrally processed on large scale, consumed by most households in West African countries (even rural, poor households), and consumed by most members of the household in relatively constant amounts. However, several important research questions remain regarding whether the use of fortified bouillon would be feasible and effective for preventing or reducing micronutrient deficiencies in communities where such deficiencies are common. Specifically, no studies have assessed the impacts of multiple micronutrient-fortified bouillon on micronutrient status. The West Africa Condiment Micronutrient Innovation Trial (CoMIT) Project aims to address this gap, to inform future discussions around fortification of bouillon cubes and related products.

Objective: This study aims to assess the impacts of household use of multiple micronutrient-fortified bouillon cubes (containing iodine in addition to vitamin A, folic acid, vitamin B12, iron, and zinc), compared to control bouillon cubes fortified with iodine only, on:

1. Micronutrient status among women 15-49 years of age and children 2-5 years of age after 9 months of intervention
2. Hemoglobin concentrations among women 15-49 years of age and children 2-5 years of age after 9 months of intervention
3. Breast milk micronutrient concentrations among lactating women 4-18 months postpartum after 3 months of intervention

Methods: This randomized, controlled doubly-masked trial will be conducted in the Kumbungu and Tolon districts in the Northern Region of Ghana, where prior data indicate that deficiencies in the selected nutrients are common. Potential participants will be: 1) non-pregnant non-lactating women of reproductive age (15 - 49 years old), 2) children 2-5 years of age, and 3) non-pregnant lactating women 4-18 months postpartum. Eligible participants will be randomly assigned to receive household rations of one of two types of bouillon cubes:

1. a multiple micronutrient-fortified bouillon cube containing vitamin A, folic acid, vitamin B12, iron, zinc, and iodine, or
2. a control cube containing iodine only

Each participant's household will receive a specific amount of bouillon cube every 2 weeks, and households will be advised to prepare their meals as usual, using the study-provided cubes. The trial duration will be 9 months (38 weeks) for non-pregnant, non-lactating women and children 2-5 years of age, and 3 months (12 weeks) for lactating women. The primary outcomes will be changes from baseline to endline in concentrations of haemoglobin and biomarkers of micronutrient status. Secondary outcomes will include change in prevalence of anaemia and micronutrient deficiency; dietary intake of bouillon and micronutrients; inflammation, malaria, and morbidity symptoms; and children's anthropometric measures and child development.

ELIGIBILITY:
Inclusion/exclusion criteria at recruitment (home visit):

Household

Inclusion criteria:

- Head of household provides oral consent for the participation of household members (index participants), and willingness to have study-provided bouillon cubes used in their household for the next 10 months.

Exclusion criteria:

* Reported chronic medical condition requiring frequent blood transfusion (e.g. severe forms of thalassemia) among any household members;
* Current participation of any household member in a clinical trial;
* Reported shrimp, wheat, milk, soy, eggs, celery, fish, or mollusk allergy, or a previous adverse reaction to bouillon by the participant or any member of their household.

Non-pregnant, non-lactating women of reproductive age

Inclusion criteria:

* Non-pregnant non-lactating women of reproductive age (15 - 49 years);
* Signed the informed consent form (or in the case of adolescents 15-17 years of age, unmarried and still living with their parents, assent provided from the index participant and consent from a parent or guardian) ;
* Planning to remain in the study area for the next 10 months;
* Willing to use study-provided bouillon in household cooking for the next 10 months;
* Not planning to become pregnant during the next 10 months.

Exclusion criteria:

* Severe illness warranting immediate hospital referral;
* COVID-19 diagnosis or exposure in the previous two weeks [individual may repeat eligibility assessment after deferral];
* Presence of morbidity symptoms suggesting COVID-19 infection (fever [temperature > 38°C], chills/shaking, dry cough, shortness of breath or difficulty breathing, loss of smell or taste within the past 72 hours) [individual may repeat eligibility assessment after deferral];
* Chronic severe medical condition (e.g. malignancy) or congenital anomalies requiring frequent medical attention or potentially interfering with nutritional status;
* Unable to provide informed consent due to impaired decision-making abilities.

Children 2-5 years of age (24-59 mo)

Inclusion criteria:

* Child 2-5 years of age (24-59 mo);
* Signed informed consent for the child's participation from a parent or guardian;
* Planning to remain in the study area for the next 10 months;
* Caregiver willing to use study-provided bouillon in household cooking for the next 10 months.

Exclusion criteria:

* Severe illness warranting immediate hospital referral;
* COVID-19 diagnosis or exposure in the previous two weeks [individual may repeat eligibility assessment after deferral];
* Presence of morbidity symptoms suggesting COVID-19 infection (fever, [temperature > 38°C], chills/shaking, dry cough, shortness of breath or difficulty breathing, loss of smell or taste within the past 72 hours) [individual may repeat eligibility assessment after deferral];
* Mid-upper arm circumference < 11.5 cm;
* Chronic severe medical condition (e.g. malignancy) or congenital anomalies requiring frequent medical attention or potentially interfering with nutritional status.

Lactating women

Inclusion criteria:

* Non-pregnant women of reproductive age (15 - 49 years), currently breastfeeding a child who is 4-18 months of age;
* Signed the informed consent form (or in the case of adolescents 15-17 years of age, unmarried and still living with their parents, provide assent from the index participant and consent from a parent or guardian);
* Planning to remain in the study area for the next 4 months;
* Planning to breastfeed for the next 4 months;
* Willing to use study-provided bouillon in household cooking for the next 4 months;
* Not planning to become pregnant during the next 4 months.

Exclusion criteria:

* Pregnancy (determined by self-report);
* Severe illness warranting immediate hospital referral;
* COVID-19 diagnosis or exposure in the previous two weeks [individual may repeat eligibility assessment after deferral];
* Presence of morbidity symptoms suggesting COVID-19 infection (fever[temperature > 38°C], chills/shaking, dry cough, shortness of breath or difficulty breathing, loss of smell or taste within the past 72 hours) [individual may repeat eligibility assessment after deferral];
* Chronic severe medical condition (e.g. malignancy) or congenital anomalies requiring frequent medical attention or potentially interfering with nutritional status;
* Unable to provide informed consent due to impaired decision-making abilities.

Exclusion criteria at screening visit for vitamin A isotope dose (WRA only):

Non-pregnant, non-lactating women of reproductive age

* Hemoglobin < 80 g/L at baseline screening visit;
* Severe illness warranting immediate hospital referral;
* COVID-19 diagnosis or exposure in the previous two weeks [individual may repeat eligibility assessment after deferral];
* Presence of morbidity symptoms suggesting COVID-19 infection (fever [temperature > 38°C], chills/shaking, dry cough, shortness of breath or difficulty breathing, loss of smell or taste within the past 72 hours) [individual may repeat eligibility assessment after deferral];
* Recent diarrhea [≥3 liquid or semiliquid stools in 72 hours]) [individual may repeat eligibility assessment after deferral];
* Reported consumption of vitamin A-rich foods (e.g., liver) in the previous 24 hours [individual may repeat eligibility assessment after deferral];
* Pregnancy (as ascertained via urine pregnancy test for human chorionic gonadotropin on the day of isotope dosing);
* Incomplete consumption of vitamin A isotope dose;
* Positive malaria RDT on the day of isotope dosing [individual may repeat eligibility assessment after deferral];
* CRP > 5 mg/L on the day of isotope dosing [individual may repeat eligibility assessment after deferral].

Exclusion criteria at baseline visit:

Non-pregnant, non-lactating women of reproductive age

* Hemoglobin < 80 g/L;
* Severe illness warranting immediate hospital referral;
* COVID-19 diagnosis or exposure in the previous two weeks [individual may repeat eligibility assessment after deferral];
* Presence of morbidity symptoms suggesting COVID-19 infection (fever [temperature > 38°C], chills/shaking, dry cough, shortness of breath or difficulty breathing, loss of smell or taste within the past 72 hours) [individual may repeat eligibility assessment after deferral];
* Pregnancy (determined by self-report).

Children 2-5 years of age

* Hemoglobin < 70 g/L;
* Severe illness warranting immediate hospital referral;
* COVID-19 diagnosis or exposure in the previous two weeks [individual may repeat eligibility assessment after deferral];
* Presence of morbidity symptoms suggesting COVID-19 infection (fever [temperature > 38°C], chills/shaking, dry cough, shortness of breath or difficulty breathing, loss of smell or taste within the past 72 hours) [individual may repeat eligibility assessment after referral];
* Severe acute malnutrition at baseline (weight-for-height Z-score < -3 SD or bilateral oedema).

Lactating women

* Severe illness warranting immediate hospital referral;
* COVID-19 diagnosis or exposure in the previous two weeks [individual may repeat eligibility assessment after deferral];
* Presence of morbidity symptoms suggesting COVID-19 infection (fever [temperature > 38°C], chills/shaking, dry cough, shortness of breath or difficulty breathing, or loss of taste or smell within the past 72 hours) [individual may repeat eligibility assessment after deferral];
* Pregnancy (determined by self-report);
* Cessation of lactation, or planning to discontinue breastfeeding in the next three months.

Exclusion criteria during course of the intervention:

Non-pregnant, non-lactating women of reproductive age

* Pregnancy (determined by self-report);
* Pregnancy (as ascertained via urine pregnancy test for human chorionic gonadotropin at pre-endline isotope dosing).

Lactating women

* Cessation of lactation (determined by self-report);
* Pregnancy (determined by self-report).

Ages: 2 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2372 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Change in vitamin A status among non-pregnant, non-lactating women | 38 weeks
  Total body vitamin A stores and estimated liver vitamin A concentration measured by retinol isotope dilution at baseline and endline
Change in vitamin A status among children 2-5 years | 38 weeks
  Plasma retinol-binding protein (RBP) concentrations, measured at baseline and endline
Change in vitamin A status among lactating women 4-18 mo postpartum | 12 weeks
  Breast milk vitamin A concentration and vitamin A per gram fat, measured at baseline and endline
Change in iron status among non-pregnant, non-lactating women | 38 weeks
  Plasma ferritin and soluble transferrin receptor concentrations, and calculated total body iron stores (BIS), measured at baseline and endline
Change in iron status among children 2-5 years | 38 weeks
  Plasma ferritin and soluble transferrin receptor concentrations, and calculated total body iron stores (BIS), measured at baseline and endline
Change in hemoglobin concentration among non-pregnant, non-lactating women | 38 weeks
  Hemoglobin concentration measured in venous blood at baseline and endline
Change in hemoglobin concentration among children 2-5 years | 38 weeks
  Hemoglobin concentration measured in venous blood at baseline and endline
Change in zinc status among non-pregnant, non-lactating women | 38 weeks
  Plasma zinc measured at baseline and endline
Change in zinc status among children 2-5 years | 38 weeks
  Plasma zinc measured at baseline and endline
Change in folate status among non-pregnant, non-lactating women | 38 weeks
  Erythrocyte folate concentrations, calculated from whole blood folate and serum folate concentrations, measured at baseline and endline
Change in folate status among children 2-5 years | 38 weeks
  Plasma folate concentrations, measured at baseline and endline
Change in vitamin B12 status among non-pregnant, non-lactating women | 38 weeks
  Plasma vitamin B12 concentrations, measured at baseline and endline
Change in vitamin B12 status among children 2-5 years | 38 weeks
  Plasma vitamin B12 concentrations, measured at baseline and endline
Change in vitamin B12 status among lactating women 4-18 months postpartum | 12 weeks
  Breast milk vitamin B12 concentrations, measured at baseline and endline

SECONDARY OUTCOMES:
Average daily household consumption of bouillon | 38 weeks
  Assessed biweekly by questionnaire, observed stocks, and wrapper counts.
Adherence to study-provided bouillon | 38 weeks
  Consumption of study-provided bouillon cubes, expressed as percentage of all bouillon consumed by the household, and as percentage of study-provided consumed by the household, assessed biweekly by questionnaire, observed stocks, and wrapper counts
Change in vitamin A status markers among non-pregnant, non-lactating women | 38 weeks
  Plasma or serum retinol and retinol-binding protein (RBP) concentrations, measured at baseline and endline
Change in serum folate concentration among non-pregnant, non-lactating women | 38 weeks
  Serum folate concentration, measured at baseline and endline
Change in plasma retinol concentration among children 2-5 years | 38 weeks
  Measured at baseline and endline
Change in iodine status among non-pregnant, non-lactating women | 38 weeks
  Urinary iodine concentration, measured at baseline and endline
Change in iodine status among children 2-5 years | 38 weeks
  Urinary iodine concentration, measured at baseline and endline
Change in iodine status among lactating women 4-18 months postpartum | 12 weeks
  Urinary iodine concentration, measured at baseline and endline
Change in urinary sodium concentrations among non-pregnant, non-lactating women | 38 weeks
  Urinary sodium concentration, expressed as sodium:potassium ratio, measured at baseline and endline
Change in inflammation among non-pregnant, non-lactating women | 38 weeks
  Plasma concentrations of acute phase proteins, measured at baseline and endline
Change in inflammation among children 2-5 years | 38 weeks
  Plasma concentrations of acute phase proteins, measured at baseline and endline
Change in current or recent malaria among non-pregnant, non-lactating women | 38 weeks
  Assessed by rapid diagnostic test at baseline and endline
Change in current or recent malaria among children 2-5 years | 38 weeks
  Assessed by rapid diagnostic test at baseline and endline
Morbidity among non-pregnant, non-lactating women | 38 weeks
  Cumulative days of symptoms over the study period, assessed by questionnaires administered biweekly
Morbidity among children 2-5 years | 38 weeks
  Cumulative days of symptoms over the study period, assessed by questionnaires administered biweekly
Morbidity among lactating women 4-18 months postpartum | 12 weeks
  Cumulative days of symptoms over the study period, assessed by questionnaires administered biweekly
Change in dietary intake among non-pregnant, non-lactating women | 38 weeks
  Dietary intake of bouillon, salt, fortifiable foods, energy, macronutrients, and micronutrients, assessed by repeated 24-hour dietary recalls at baseline and endline
Change in dietary intake among children 2-5 years | 38 weeks
  Dietary intake of bouillon, salt, fortifiable foods, energy, macronutrients, and micronutrients, assessed by repeated 24-hour dietary recalls at baseline and endline
Dietary intake among lactating women 4-18 months postpartum | 4 weeks
  Dietary intake of bouillon, salt, fortifiable foods, energy, macronutrients, and micronutrients, assessed by repeated 24-hour dietary recalls at baseline
Change in anemia among non-pregnant, non-lactating women | 38 weeks
  Hemoglobin concentrations < 12 g/dL, measured at baseline and endline
Change in anemia among children 2-5 years | 38 weeks
  Hemoglobin concentrations < 11 g/dL, measured at baseline and endline
Change in micronutrient deficiency among non-pregnant, non-lactating women | 38 weeks
  Based on biomarkers of micronutrient status (vitamin A, iron, zinc, folate, vitamin B12), measured at baseline and endline
Change in micronutrient deficiency among children 2-5 years | 38 weeks
  Based on biomarkers of micronutrient status (vitamin A, iron, zinc, folate, vitamin B12), measured at baseline and endline
Change in low milk nutrient concentrations among lactating women 4-18 months postpartum | 12 weeks
  Based on concentrations of vitamin A and vitamin B12, measured at baseline and endline
Systolic and diastolic blood pressure among non-pregnant, non-lactating women | 38 weeks
  Assessed by portable device
Hypertension among non-pregnant, non-lactating women | 38 weeks
  Based on blood pressure measured by portable device
Change in faecal calprotectin concentrations among children 2-5 years | 38 weeks
  Stool samples collected at baseline and endline
Change in height-for-age Z score and stunting (HAZ < -2) among children 2-5 years | 38 weeks
  Standing height, standardized using WHO child growth standards
Change in weight-for-height Z score and wasting (WHZ < -2) among children 2-5 years | 38 weeks
  Standardized using WHO child growth standards
Change in cognitive development among children 2-5 years | 38 weeks
  Malawi Developmental Assessment Tool (MDAT) scores in 4 domains (gross motor, fine motor, language, social)
Fecal microbiota among children 2-5 years | 38 weeks
  Stool samples collected at baseline and endline
Change in cognitive development among children 2-5 years | 38 weeks
  Early Years Toolbox scores at baseline and endline

OTHER OUTCOMES:
Household food security | 38 weeks
  Assessed monthly using the Household Food Insecurity and Access Scale (HFIAS)
Household water security | 38 weeks
  Assessed monthly by the Household Water Insecurity Experience Scale (HWISE)
Change in weight-for-age Z score and underweight (WAZ < -2) among children 2-5 years | 38 weeks
  Standardized using WHO child growth standards
Change in zinc protoporphyrin (ZPP) concentrations | 38 weeks
  Measured by portable device

CONTACTS AND LOCATIONS:
Overall Officials: Reina Engle-Stone, PhD, Principal Investigator — Department of Nutrition, UC Davis; Seth Adu-Afarwuah, PhD, Principal Investigator — University of Ghana
Locations (1):
- University of Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will commit to Global Access. The investigators intend to 1) publish journal articles describing the study results with an Open Access license, 2) make available information about study methods, such as protocols or standard operating procedures, on the study website, and 3) make available de-identified datasets upon request by the study sponsor or other investigators. Material/DataTransfer Agreements will be developed between study collaborators, sponsor, and any organizations that may request the data; terms of the agreement will be subject to the data handling and storage procedures approved by the University of California, Davis Institutional Review Board (IRB) and Ghana Health Services Ethical Review Committee (GHS-ERC). Organizations that may request the data; terms of the agreement will be subject to the data handling and storage procedures approved by the University of California, Davis IRB and GHS-ERC.

REFERENCES:
- [Derived] Engle-Stone R, Wessells KR, Haskell MJ, Kumordzie SM, Arnold CD, Davis JN, Becher ER, Fuseini AD, Nyaaba KW, Tan X, Adams KP, Lietz G, Vosti SA, Adu-Afarwuah S. Effect of multiple micronutrient-fortified bouillon on micronutrient status among women and children in the Northern Region of Ghana: Protocol for the Condiment Micronutrient Innovation Trial (CoMIT), a community-based randomized controlled trial. PLoS One. 2024 May 6;19(5):e0302968. doi: 10.1371/journal.pone.0302968. eCollection 2024. PMID 38709803